CLINICAL TRIAL: NCT03290976
Title: Impact of Integrative Medicine on Chemotherapy-Induced Peripheral Neuropathy: A Multi-centered, Randomized Controlled Trial
Brief Title: Integrative Medicine for Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Chaim Sheba Medical Center (Other)
Collaborators: Bnai Zion Medical Center (Other Government); Lin Medical Center, Haifa (Other); Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Noah Samuels, Medical Director, Tal Center for Integrative Oncology, Institute of Oncology, The Chaim Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4462-17-SMC
Record Dates: First submitted 2017-09-13; First posted 2017-09-25 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Patient-preference, randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The control group will consist of patients who choose not to undergo CIM treatments for their CIPN-related symptoms. Participants in this arm of the study will receive standard conventional supportive care, as provided by their oncology health care professionals (HCPs), and closely monitored for any changes in the severity of their CIPN-related symptoms.
- Intervention Group A: Single Modality (acupuncture) (Active Comparator): Patients choosing to undergo CIM treatments, in addition to standard conventional care: Acupuncture x2/week, for 6 weeks.
  Interventions: Other: Acupuncture
- Intervention Group B: Multi-modality (acupuncture "plus") (Active Comparator): Patients choosing to undergo CIM treatments, in addition to standard conventional care: Acupuncture with additional CIM treatment modalities, x2/week, for 6 weeks.
  Interventions: Other: Acupuncture; Other: Multi-modality (Acupuncture "plus")

INTERVENTIONS:
Other: Acupuncture — Acupuncture treatments will be patient-tailored, with the acupuncture points (acu-points) to be selected by the acupuncturist at each treatment session, in accordance with the dynamic of the patient's symptoms, concerns and expectations. At the same time, acupuncturists will be required to choose at least 5 of the following 11 acupoints, which are to be incorporated into their treatment regimen:
  Lower limb points: Liver (LIV) 3, Spleen (SP) 4, SP6, Stomach (ST) 36, Gallbladder (GB) 34, Kidney (KID) 3, LIV8, Web (Bafeng) points Upper limb points: Large Intestine (LI) 4, LI 11, LI10, Pericardium (PC) 6, Triple Warmer (TW) 3/4/5
  Arms: Intervention Group A: Single Modality (acupuncture); Intervention Group B: Multi-modality (acupuncture "plus")
Other: Multi-modality (Acupuncture "plus") — A number of additional CIM treatment modalities will be added to the acupuncture treatment in this arm of the study, in accordance with the practitioners available at each of the participating study centers. These will include one of more of the following:
  * Manual-movement therapies - e.g. acupressure/reflexology, self- and caregiver-practiced acupressure
  * Mind-body therapies - e.g. relaxation/imagery method, Anthroposophic music therapy The multimodal CIM treatment regimen will be re-evaluated at each session, and adapted according to the concerns and expectations of the patients, as well as the recommendation of the treating CIM practitioner.
  Arms: Intervention Group B: Multi-modality (acupuncture "plus")

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common and often debilitating complication of cancer treatments. There is presently no known treatment which can prevent the onset of CIPN, with treatment of existing symptoms limited to reducing the dose intensity of the offending agent. Clinical research has shown that complementary/integrative medicine (CIM) modalities such as acupuncture and reflexology may be effective in relieving CIPN-related symptoms. The present study will included 120 patients suffering from CIPN-related symptoms, and will take place at 3 medical centers in Israel which provide CIM treatments to oncology and hemato-oncology patients. Participants will be allocated to either the control arm (standard conventional supportive care; n=40) or to the intervention arm of the study (standard care with CIM treatments; n=80), based on their preference. Patients in the treatment arm of the study will be randomly allocated to either twice-weekly, single modality acupuncture treatments (n=40), or to a multi-modality treatment program (n=40), which will include acupuncture and additional CIM modalities (i.e., manual-movement and mind-body therapies), for a 6-week period.

The effect of CIM treatments in reducing the severity of CIPN-related symptoms will be assessed at baseline and at 6- and 9-week follow-up visits, using the Functional Assessment of Cancer Therapy -Taxane (FACT-Tax) tool; the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - C30 (EORTC QLQ-C30); and the Measure Yourself Concerns and Well-being (MYCAW) questionnaire. Interim assessment of symptom severity will be conducted by the study nurse throughout the study period, through either telephone or e-mail. Additional study outcomes will include the safety of the CIM treatments; QOL-related concerns which may affect CIPN-related symptoms (e.g., anxiety, depression, sleep disturbances, etc.), as well as issues related to body image and coping with CIPN; physiological assessment of CIPN using a von Frey test (with hairs of varying diameters to assess the threshold for touch evoked sensations); and adherence to the planned oncology treatment regimen, as measured by the Relative Dose Intensity (RDI) calculation.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with breast or gynecological cancers who are undergoing a treatment regimen which includes taxane-based chemotherapy (e.g., Paclitaxel, Docetaxel); or
* Patients of either gender with hematological malignancies who are undergoing a treatment regimen which includes neuropathy-inducing agents (e.g., bortezumab for multiple myeloma, etc.).
* Eligible patients will report altered sensations and/or pain in the areas of the feet and or hands, with a score of ≥ 2 (moderate-to-severe) for chemotherapy-induced peripheral neuropathy on the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events - version 4.0 (CTC-AE.v-4.0)
* The onset of CIPN-related symptoms must be recent, following a recently-administered course of chemotherapy and with symptoms appearing no more than a month prior to study recruitment.

Patients must be able to comply with the study protocol, which includes weekly follow-up visits, either in person or by phone; completion of the study questionnaires, in accordance with the study protocol; and, for patients in the treatment arm of the study, attending twice-weekly CIM treatment sessions.

Exclusion Criteria:

- Patients not fulfilling the inclusion criteria, or those with a history of chronic medical conditions which predispose to the development of CIPN (e.g., diabetes mellitus, alcohol abuse), will be ineligible for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Symptom Severity(neuropathy): Functional Assessment of Cancer Therapy -Taxane (FACT-Tax) tool | Up to 9 weeks
  CIPN-related symptoms
Symptom Severity(neuropathy): European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Up to 9 weeks
  CIPN-related symptoms
Symptom Severity(neuropathy): Measure Yourself Concerns and Well-being (MYCAW) questionnaire: | Up to 9 weeks
  CIPN-related symptoms

SECONDARY OUTCOMES:
Symptom Severity(additional concerns): Functional Assessment of Cancer Therapy -Taxane (FACT-Tax) tool | Up to 9 weeks
  Additional QOL-related concerns
Symptom Severity(additional concerns): European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Up to 9 weeks
  Additional QOL-related concerns
Symptom Severity(additional concerns): Measure Yourself Concerns and Well-being (MYCAW) questionnaire: | Up to 9 weeks
  Additional QOL-related concerns
Symptom Severity(neuropathy): Physiological Assessment of CIPN Severity | Up to 9 weeks
  The von Frey test (Semmes Weinstein Monofilament Set, Bioseb In Vivo Research Instruments, France/USA).
Adherence to Chemotherapy Regimen: Relative Dose Intensity (RDI) | After 9 weeks
  RDI = Dose Administered (mg) / Interval between treatments (days) ÷ Planned Dose (mg) / Planned Interval between treatments (days)
Adverse Effects Associated with CIM treatments | After 9 weeks
  Registering of any adverse events believed to be related to the study intervention treatments

CONTACTS AND LOCATIONS:
Overall Officials: Elad Schiff, MD, Principal Investigator — Bnai Zion Medical Center, Haifa; Eran Ben-Arye, MD, Principal Investigator — Lin Medical Center, Haifa
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ben-Arye E, Gamus D, Samuels N, Schiff E, Hausner D, Gressel O, Attias S, Lavie O, David A, Shulman K, Agbarya A. Acupuncture and integrative oncology for taxane-induced peripheral neuropathy: a randomized multicentered study. Int J Gynecol Cancer. 2023 May 1;33(5):792-801. doi: 10.1136/ijgc-2022-004004. PMID 36600535